CLINICAL TRIAL: NCT02779608
Title: The Study of Intraperitoneal Docetaxel Plus S-1 for Malignant Ascites Due to Far Advanced Gastric Cancer
Brief Title: The Study of Intraperitoneal Docetaxel Plus S-1 for Malignant Ascites
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, luo fen, Professor in general surgery, Huashan hospital Fudan University, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ifen
Record Dates: First submitted 2016-05-15; First posted 2016-05-20 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Stomach Neoplasms; Peritoneal Metastasis
Keywords: malignant ascites
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; S 1 (combination); Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraperitoneal docetaxel and oral S-1 (Experimental): Docetaxel is diluted in 1litre normal saline and administered intraperitoneal（IP）at a dose of 60 mg/m2 over 1 hour on day 1. S-1 was administered orally twice daily at a dose of 40mg/m2 per day for 14 consecutive days, followed by 7 days of rest.
  Intervention: Drug: Intraperitoneal docetaxel Intervention：Drug：Oral S-1
  Interventions: Drug: intraperitoneal docetaxel; Drug: oral S-1

INTERVENTIONS:
Drug: intraperitoneal docetaxel — One peritoneal access port will be implanted in subcutaneous space of patients' abdominal wall after laparoscopic exploration.Then intraperitoneal docetaxel in 1litre normal saline will be administered through the port
  Other Names: intraperitoneal chemotherapy
Drug: oral S-1 — 40mg/m² twice daily on day 1-14 every 3 weeks
  Other Names: systemic chemotherapy

SUMMARY:
This is a clinical Study to evaluate the effect, survival benefit and safety of intraperitoneal docetaxel combined with oral S-1 for advanced gastric cancer with malignant ascites.

DETAILED DESCRIPTION:
Peritoneal metastasis(PM) is common in advanced gastric cancer and associated with a poor prognosis. The median survival time is 3 to 4 months and even shorter in the patients with malignant ascites. Systemic chemotherapy is considered to be less effective against peritoneal metastasis (PM) due to the existence of the blood-peritoneal barrier (BPB), which inhibits the movement of drugs from systemic circulation to the peritoneal cavity.

S-1 is one kind of oral fluoropyrimidine derivatives and has been reported to be effective on PM. Docetaxel (DTX) has a pharmacokinetic advantage after intraperitoneal（IP）delivery which is hundreds of times higher than systemic administration. The use of S-1 and docetaxel has been studied in some phase II trials. Fujiwara and Fushida reported the usefulness of IP docetaxel combined with oral S-1 regimen in gastric cancer with PM respectively，the median survival time can exceed 16 months and one year survival rate was over 70%. Therefore, the investigators suppose IP docetaxel and oral S-1 can also be effective for gastric cancer with malignant ascites and start this study.

This is a single center, open-label, prospective clinical trial. Patients with histological proven gastric cancer with ascites, who fulfill the inclusion and exclusion criteria, can be recruited in this study. Patients will be firstly received laparoscopic exploration for Peritoneal Cancer Index (PCI）score, extraction of 100ml ascites for cytology examination, and one peritoneal access port is implanted in the subcutaneous space of the lower abdomen. Then patients were treated with chemotherapy on the first day after operation, the regimen as follows: DTX is administered IP at a dose of 60 mg/m2 on day 1. DTX is diluted in 1 litre normal saline and administered through the implanted peritoneal access port over 1 hour. S-1 was administered orally twice daily at a dose of 80 mg/m2 per day for 14 consecutive days, followed by 7 days of rest. The treatment course will be repeated every three weeks until observation of disease progression or unacceptable toxicity. Before each intraperitoneal chemotherapy, investigators extract 50-100 ml ascites for cytology pathologic examination, the abdominal CT will be reviewed after every three course to evaluate the volume of ascites.

The volume of ascites before and after therapy, PCI scores, ascites cytology results, complications, side effects and conditions of survival state and follow-up will be recorded and analyzed to evaluate the effect, survival benefit and safety of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-75years
2. Histologic confirmation of gastric adenocarcinoma
3. Positive peritoneal cytology or histological proven PM
4. Ascites in CT scan
5. Performance status (PS) ≤ 2 on Eastern Cooperative Oncology Group (ECOG) scale
6. Adequate bone marrow and organ functions as defined below:

   Leucocyte≥3,000/ul Absolute neutrophil counts ≥1,500/uL Platelet≥100,000/uL Total bilirubin≤1.5mg/dl ALT，AST≤ 2x ULN serum creatinine ≤1.5mg/dl
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
8. Provision of written informed consent

Exclusion Criteria:

1. Presence of non-curable factors such as distant metastasis to liver or lung except of peritoneum
2. Other severe medical conditions such as symptomatic infectious disease,active hemorrhage/bleeding, or obstructive bowel disease
3. Life expectation ≤ 3 months
4. With other malignant tumor
5. allergy to therapeutic drugs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
response rate of ascites | 9 weeks
  From date of enrollment to three cycles of treatment，the ascites is evaluated by the Japanese conventional five-point method

SECONDARY OUTCOMES:
one year survival rate | 1 year
  From date of enrollment until 1 year
side effects of chemotherapy | 1 week to 18 weeks
  Grade refers to Common Terminology Criteria for Adverse Events（CTCAE）Version4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes